CLINICAL TRIAL: NCT07393373
Title: Phase 2, Open-Label, Long-Term, Extension (OLE) Study of Infigratinib, an FGFR 1-3-Selective Tyrosine Kinase Inhibitor, in Children With Hypochondroplasia: ACCEL OLE
Brief Title: Open-Label, Long-Term, Extension Study of Infigratinib in Children With Hypochondroplasia
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: QED Therapeutics, a BridgeBio company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QBGJ398-205
Record Dates: First submitted 2026-01-19; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Hypochondroplasia
Keywords: skeletal dysplasia; endochondral ossification; hypochondroplasia; HCH; shortened proximal limbs; fibroblast growth factor receptor 3; FGFR3; endochondral bone formation; disproportionate short stature; quality of life; dwarfism; bone diseases; musculoskeletal diseases; osteochondrodysplasia; functional abilities; annualized growth velocity; annualized height velocity; growth; genetic diseases; congenital; AHV; AGV; Pathogenic variants
MeSH Terms: conditions — Hypochondroplasia; Mucopolysaccharidosis IV; Dwarfism; Bone Diseases; Musculoskeletal Diseases; Osteochondrodysplasias; Genetic Diseases, Inborn | interventions — infigratinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1: Rollover subjects (Experimental): Children who have completed QED-sponsored interventional study with infigratinib
  Interventions: Drug: Infigratinib

INTERVENTIONS:
Drug: Infigratinib — Infigratinib to be administered by mouth and initiated at the last dose level received in the ACCEL 2/3 study or at the dose selected to be further evaluated after proof-of-concept is established for Phase 2 portion of ACCEL 2/3.

SUMMARY:
Phase 2, multicenter, OLE study to evaluate the long-term safety, tolerability, and efficacy of infigratinib, an FGFR (fibroblast growth factor receptor) 1-3-selective tyrosine kinase inhibitor, in participants with Hypochondroplasia (HCH) who previously completed ACCEL 2/3, and potentially additional participants who completed ACCEL. Participants rolling over directly from the observational ACCEL study must have had at least a 6-month period of growth assessment in that study.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria for Participants Rolling Over from ACCEL 2/3

  1. Pediatric participants with HCH who have completed ACCEL 2/3
  2. Negative pregnancy test in girls ≥10 years of age or girls of any age who have experienced menarche

Exclusion Criteria:

* Exclusion Criteria for Participants Rolling Over from ACCEL 2/3

  1. Participant has concurrent medical condition that, in the view of the PI and/or sponsor, would interfere with study participation or safety evaluations
  2. Participants who developed a medical condition that requires the initiation of treatment with a prohibited medication
  3. Participants who prematurely discontinued ACCEL 2/3
  4. Participants who have reached final height or near final height
  5. Current participation in an ongoing clinical study with a sponsor other than QED

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 135 (Estimated)
Dates: Start 2026-04-21 (Estimated); Primary Completion 2036-05-31 (Estimated); Study Completion 2036-05-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events (TEAE) and serious TEAE | 10 years
Changes over time in standing height Z-score in relation to HCH and non-HCH growth charts | 10 years

SECONDARY OUTCOMES:
Changes over time in AHV Z-score | 10 years
Changes over time in body proportions | 10 years
Changes over time in weight Z-score | 10 years
Changes overtime in BMI | 10 years
Age of puberty onset and time to Tanner stage ≥4 | 10 years
Changes over time in body composition as assessed by DXA (dual x-ray absorptiometry) scans | 10 years
Changes over time in bone morphology/density by x-ray and DXA | 10 years
Change in psychomotor function assessed by age-appropriate computerized tests (Detection Test) | 10 years
Change in attention assessed by age-appropriate computerized tests (Identification Test) | 10 years
Change in visual learning assessed by age-appropriate computerized tests (One Card Learning Test) | 10 years
Change in working memory assessed by age-appropriate computerized tests (One Back Test) | 10 years
Changes over time in severity of epilepsy measured by frequency and adverse event grading | 10 years
Changes in health-related Quality of life [HRQoL] as assessed by Pediatric Quality of Life Inventory (PedsQL) | 10 years
Changes in health-related Quality of life [HRQoL] as assessed by Quality of Life in Short Stature Youth questionnaire (QoLISSY) | 10 years
Severity of the physical functioning challenges as assessed by Patient/Parent Global Impression of Severity (PGI-S) | 10 years
Severity of the physical functioning challenges as assessed by Patient/Parent Global Impression of Change (PGI-C) | 10 years
Subject and caregiver evaluation of treatment benefit as assessed by a qualitative interview | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: QED Therapeutics SVP, Clinical Development, Study Director — QED Therapeutics, a BridgeBio company
Locations (25):
- United States (8):
  - UCSF Benioff Children's Hospital, Oakland, California
  - Childrens Hospital Colorado, Aurora, Colorado
  - Children's National Hospital, Washington D.C., District of Columbia
  - Johns Hopkins School of Medicine, Baltimore, Maryland
  - University of Missouri, Columbia, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Wisconsin Madison - Waisman Center Bone Dysplasia Clinic, Madison, Wisconsin
- Murdoch Children's Research Institute, Parkville, Victoria, Australia
- Canada (3):
  - London Health Sciences Centre - Children's Hospital of Western Ontario, London, Ontario
  - Children's Hospital of Eastern Ontario Research Institute, Ottawa, Ontario
  - Université de Montréal - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
- France (3):
  - Hôpital Femme Mère Enfant, Bron
  - Hôpital Universitaire Necker-Enfants Malades, Paris
  - Centre Hospitalier Universitaire (CHU) de Toulouse - Hôpital des Enfants, Toulouse
- Norway (2):
  - Haukeland University Hospital, Bergen
  - Paediatric Clinical Research Unit at Osla University Hospital, Oslo
- Hospital Pediátrico de Coimbra, Coimbra, Portugal
- KK Women's and Children's Hospital, Singapore, Singapore
- UCA Hospital MiKS, Vitoria-Gasteiz, Spain
- Astrid Lindgren Children's Hospital, Solna, Sweden
- United Kingdom (4):
  - The Portland Hospital for Women and Children, London, England
  - Manchester University, Manchester, England
  - Sheffield Children's Hospital, Sheffield, England
  - Glasgow Clinical Research Facility, Queen Elizabeth University Hospital, Glasgow, Scotland

IPD SHARING:
Plan to Share IPD: No